CLINICAL TRIAL: NCT07100028
Title: Comparison of Hall Technique vs Conventional Technique in Permanent Teeth
Brief Title: Hall Technique vs Conventional Technique in Permanent Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, GIZEM ERBAS UNVERDI, Assistant prof, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Hall technique-permanent
Record Dates: First submitted 2025-06-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dental Caries; Crowned Posterior Teeth
Keywords: hall technique; permanent teeth; crown
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Two technique on two molars in one patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSC crown with conventional technique (Active Comparator): SSC crown placement using conventional technique
  Interventions: Other: SSC crown with Hall technique
- SSC crown with Hall technique (Experimental): SSC crown placement using Hall technique
  Interventions: Other: SSC with conventional technique

INTERVENTIONS:
Other: SSC crown with Hall technique — SSC crown placement using Hall technique
  Arms: SSC crown with conventional technique
Other: SSC with conventional technique — SSC placement using conventional technique
  Arms: SSC crown with Hall technique

SUMMARY:
The purpose of this study is to evaluate and compare the clinical and radiological performance of stainless steel crowns using conventional and Hall technique on permanent molars

DETAILED DESCRIPTION:
Stainless Steel Crowns will be applied on two permanent molar teeth in a split mouth design. 96 patients will be included in the study. The teeth will be randomized into two groups according to the applying methods: 1) Traditional method 2) Hall technique.

Oral hygiene index (Green & Vermillion), Plaque index (Sillness & Löe), gingival health (Löe & Sillness), level of gingival margin, crown retention and success, wear, occlusion, clinical pulpal health (spontaneous pain, mucosal swelling/fistula presence, mobility, percussion/palpation tenderness) and radiographic pulpal health (periradicular/interradicular radiolucency, lamina dura loss, internal/external root resorption, pulp canal obliteration) will be evaluated and photographic records will be taken.

The evaluation of the restorations will be performed at baseline, and 1., 3., 6., 12., 18., 24. months. The measurement of vertical hight on occlusion will be performed before and immediate after the treatment, at 2 weeks and 1., 2. and 3.months.

Fisher's Exact test, Kaplan-Meier Survival Curves, Log-rank test, Mann Whitney U test, and Friedman test will be performed for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The child volunteers and their parents who read and agreed to the informed consent form.
2. The presence of excessive loss of material or extensive enamel defects in at least two permanent molars that require crown application.
3. The presence of antagonist teeth of the teeth to be crowned.
4. All treatments on the patient's other teeth have been completed.
5. The patient who does not have temporomandibular joint (TMJ) problems.
6. Children who have cooperation to allow the dental procedure to be completed.

Exclusion Criteria:

1. Child volunteers or parents who refuse to participate in the study.
2. The patient who has a chronic disease.
3. Patients undergoing orthodontic treatment
4. The patient has missing teeth on the treated side.
5. The need for vital or non-vital pulp treatment of the tooth.
6. The child volunteers and their parents did not accept the aesthetic appearance of the stainless steel crown.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiological performance of SSCs placed with Hall of conventional technique | 2 years
  The primary outcome 'success' was defined as the "absence of major failure," a measure encompassing clinical and radiographic signs of irreversible pulpitis or infectious complications (spontaneous pain, pulp infection, or periradicular pathology, loss of lamina dura on radiographs).

SECONDARY OUTCOMES:
Clinical measurements of SSCs placed with Hall of conventional technique | 2 years
  * Plaque index (Sillness & Löe index), gingival health (Löe & Sillness index) scores will be measured.
  * Treatment longevity, will be measured as the time interval between the groups and the final follow-up date.
  * Retention of the SSC, defined as the presence or absence of SSC.
  * Normalisation time of the vertical height of the occlusion in Hall technique group.

CONTACTS AND LOCATIONS:
Overall Officials: zafer cavit cehreli, prof.dr., Study Chair
Locations (1):
- Hacettepe university, pediatric dentistry, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD is available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: IPD is available from the corresponding author on reasonable request.